CLINICAL TRIAL: NCT00956488
Title: Supported Treadmill Ambulation Training (STAT) for Patients Diagnosed With Amyotrophic Lateral Aclerosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 07-08-15E
Record Dates: First submitted 2009-08-10; First posted 2009-08-11 (Estimated); Last update posted 2022-04-21 (Actual); Status verified 2013-07

CONDITIONS: Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Lou Gehrig's Disease
Keywords: Exercise for Amyotrophic lateral sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- supported treadmill ambulation training (Experimental)
  Interventions: Behavioral: Treadmill Exercise

INTERVENTIONS:
Behavioral: Treadmill Exercise — The intervention will consist of 30 minutes of exercise, performed 3 times per week for 8 weeks (24 sessions). Patient will walk on a treadmill with up to 40% of their body weight supported by a body weight support system with an overhead harness. The training session duration will be 60 minutes consisting of six intervals of 5 minutes exercise, interspersed with 6 intervals of 5 minutes rest to avoid overwork weakness and fatigue. Five minute exercise intervals should be sufficient for patients to reach a steady state. Patients will build up their endurance to this training level at their own pace as tolerated. Walking speed will be determined as tolerated by each patient. Exercise intensity will be guided by each patient's own perception of exertion, but not to exceed level 12-13 (mild to moderate) on the modified Borg perceived exertion scale, and by oxygen saturation (Sa O2) ≥ 90% monitor by handheld pulse Oximeter.

SUMMARY:
The purpose of this study is to find out if supervised exercise training using a treadmill with partial weight support is safe and has an impact on gait and function of persons with Amyotrophic lateral sclerosis.

DETAILED DESCRIPTION:
Twenty ALS patients who are independent in their transfer with assistive devise such as walker, cane, or AFO will be offered the opportunity to participate in this study. 20 subjects will be enrolled at Carolinas ALS/Neuromuscular Center at the Carolinas HealthCare System. Eligible subjects will return for 26 sessions, each lasting between 1-2 hours. At Session 1 (4 weeks pre-treatment), assessments of muscle strength, spasticity, gait, and balance will be performed, which will take between 30-60 minutes. At Sessions 2-25, patients will do supported treadmill ambulation training at a very low speed 3 times a week for 6 weeks under the supervision of the physical therapist. Each session will have 30 minutes of direct ambulation with the suspension system and treadmill over a 60 minute period of time. Additionally, at sessions 13 and 26 (4 and 8 weeks post-treatment), the assessments of muscle strength, spasticity, gait, and balance will be repeated. Needle EMG to assess denervation potential will be performed at base line and at the conclusion of the study. The study will last a total of 26 weeks for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Clinically probable or definite diagnosis of ALS/MND
* Able to stand independently and ambulate for six minutes with their assistive devices
* Able to complete the 25 foot walk in less than 1 minute
* Vital Capacity of over 65% predicted
* 25 to 75 years of age
* Not a pregnant woman
* Able to provide informed consent and to comply with training and assessment procedures

Exclusion Criteria:

* Unstable angina or severe left main coronary disease
* End-stage congestive heart failure
* Severe valvular heart disease
* Malignant or unstable arrhythmias
* Elevated resting blood pressure (systolic, 200mmHg; diastolic, 110mmHg)
* Large or expanding aortic aneurysm
* Known cerebral aneurysm or recent intracranial bleed
* Uncontrolled or end-stage systemic disease
* Acute retinal hemorrhage or recent ophthalmologic surgery
* Acute or unstable musculoskeletal injury

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Twenty Five Foot Walk Test (25FWT) | baseline, after 4 weaks and 8 weaks post training
The Six-Minute Walk Test (6MWT) | baseline, after 4 weaks and 8 weaks post training
Fatigue severity scale (FSS) | baseline, after 4 weaks and 8 weaks post training

SECONDARY OUTCOMES:
Muscle strength | baseline, after 4 weaks and 8 weaks post training
ALS functional rating scale (ALSFRS-R) | baseline, after 4 weaks and 8 weaks post training
Vital Capacity | baseline, after 4 weaks and 8 weaks post training
Beck Depression Inventory (BDI) | baseline, after 4 weaks and 8 weaks post training

CONTACTS AND LOCATIONS:
Locations (1):
- Carolinas ALS Clinical Resarch Center, Charlotte, North Carolina, United States